CLINICAL TRIAL: NCT04906200
Title: Randomized Controlled Trial of Young, Empowered & Strong (YES), a Web-Based Patient-Reported Symptom Monitoring and Self-Management Portal for Adolescent and Young Adult Breast Cancer Survivors
Brief Title: Web-Based Symptom Monitoring and Self-Management Portal (YES) for Adolescent and Young Adult Breast Cancer Survivors
Acronym: YES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Dana-Farber Cancer Institute (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Michelle Naughton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-21035; NCI-2021-03962 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U01CA246648 (NIH)
Record Dates: First submitted 2021-05-13; First posted 2021-05-28 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC V8; Anatomic Stage I Breast Cancer AJCC V8; Anatomic Stage IA Breast Cancer AJCC V8; Anatomic Stage IB Breast Cancer AJCC V8; Anatomic Stage II Breast Cancer AJCC V8; Anatomic Stage IIA Breast Cancer AJCC V8; Anatomic Stage IIB Breast Cancer AJCC V8; Anatomic Stage III Breast Cancer AJCC V8; Anatomic Stage IIIA Breast Cancer AJCC V8; Anatomic Stage IIIB Breast Cancer AJCC V8; Anatomic Stage IIIC Breast Cancer AJCC V8; Prognostic Stage 0 Breast Cancer AJCC V8; Prognostic Stage I Breast Cancer AJCC V8; Prognostic Stage IA Breast Cancer AJCC V8; Prognostic Stage IB Breast Cancer AJCC V8; Prognostic Stage II Breast Cancer AJCC V8; Prognostic Stage IIA Breast Cancer AJCC V8; Prognostic Stage IIB Breast Cancer AJCC V8; Prognostic Stage III Breast Cancer AJCC V8; Prognostic Stage IIIA Breast Cancer AJCC V8; Prognostic Stage IIIB Breast Cancer AJCC V8; Prognostic Stage IIIC Breast Cancer AJCC V8
MeSH Terms: conditions — Breast Carcinoma In Situ | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (YES portal) (Experimental): Patients receive access to YES portal for 9 months. Patients also complete surveys at baseline and 3, 6, and 9 months.
  Interventions: Other: Internet-Based Intervention; Other: Survey Administration
- Group B (usual care) (Active Comparator): Patients receive usual care for 9 months. Patients also complete surveys at baseline and 3, 6, and 9 months. After 9 months, patients may also receive access to YES portal for 3 months.
  Interventions: Other: Best Practice; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Group B (usual care)
Other: Internet-Based Intervention — Receive access to YES portal
  Arms: Group A (YES portal)
Other: Survey Administration — Complete survey

SUMMARY:
This clinical trial compares a web-based patient-reported symptom monitoring and self management portal, the Young, Empowered & Strong (YES), to standard therapy in managing symptoms in adolescent and young adult breast cancer survivors. YES is a web-based portal (website) to help monitor issues or symptoms women with breast cancer may experience. The YES portal may improve the quality of life of young breast cancer survivors. The YES portal may help manage symptoms and provide useful information/resources.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of the YES intervention compared to usual care in improving quality of life (QOL), as measured by the Quality of Life in Adult Cancer Survivors (QLACS) at 6-months (primary outcome).

II. To determine the efficacy of the YES intervention compared to usual care in reducing specific adolescent and young adult (AYA) breast cancer (BC) concerns and symptoms at 6-months.

III. To determine the sustainability of the effects of YES on AYA concerns, symptoms, and QOL at 9 months, after the completion of the 6-month active intervention period.

EXPLORATORY OBJECTIVE:

I. To explore potential moderators and mediators of intervention efficacy, and to explore the potential effects of the intervention on inflammatory and other biomarkers including genetic profiles.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP A: Patients receive access to the YES portal for 9 months. Patients also complete surveys at baseline and 3, 6, and 9 months.

GROUP B: Patients receive usual care for 9 months. Patients also complete surveys at baseline and 3, 6, and 9 months. After 9 months, patients may also receive access to the YES portal for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 15-39 years at diagnosis of a stage 0-III breast cancer
* Within 3 years of breast cancer diagnosis
* No known evidence of breast cancer recurrence (local or distant) or second primary breast cancer
* No prior history of new other malignancy since their breast cancer diagnosis (other than non-melanoma skin cancer)
* Able to speak, understand and read English
* Cognitively able to complete the study requirements
* Ability to access medical records from treating hospital
* Willing to provide cell phone number and/or email address, and willing to receive email and/or text messages from the study team either with their own smartphone or one provided by the study team if they do not have their own to use
* Pregnant survivors are also eligible for this protocol, given that fertility and pregnancy are important AYA issues

Exclusion Criteria:

* Individuals under age 15 or over age 42
* Stage IV or metastatic breast cancer
* Males with breast cancer are not being recruited to this protocol. In the AYA age group, only a miniscule proportion of breast cancers occur in males. For this reason, the YES portal intervention materials have been targeted for young women

Ages: 15 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the Young, Empowered & Strong (YES) intervention in improving quality of life (QOL) | Up to 6 months
  Will determine the efficacy of the YES intervention compared to usual care in improving QOL, as measured by the Quality of Life in Adult Cancer Survivors Scale at 6-months (primary outcome). The QLACS contains 47 items scored on a 1 (never) to 7 (always) scale. The 47 items are grouped into 12 domains (7 generic and 5 cancer-specific). A QLACS generic summary score is calculated by adding the 7 constituent domain scores, so that a lower score (range: 31-143) corresponds to higher QOL. A QLACS cancer-specific summary score (range: 16-99) is calculated by adding the constituent domain scores of all but the "benefits" domain. The benefits domain is scored separately (range: 4-28).

SECONDARY OUTCOMES:
Efficacy of the YES intervention in reducing specific adolescent and young adult (AYA) breast confident (BC) concerns and symptoms at 6-months compared to baseline. | Up to 6 months
  AYA concerns and symptoms will be measured by items from the AYA HOPE Study questionnaire that asks patients to indicate their need for information regarding a range of AYA survivorship-focused issues, including fertility, diet and nutrition, physical activity, weight management, survivorship care, recurrence concerns, and financial support for medical care. Symptoms assessed include sexual problems, anxiety, fatigue, stress, depression, sleep problems, hot flashes, and musculoskeletal complaints. Changes in concerns and symptoms will be examined using the frequencies of the report of needs and symptoms between baseline and 6 months. Lower frequencies of concerns and symptoms, as compared to their baseline levels, both indicate better outcomes.
Sustainability of the effects of YES on AYA concerns and symptoms | Up to 9 months post-baseline, after the completion of the 6-month active intervention period
  Frequencies of AYA concerns for information and frequencies of symptoms at 9 months will be compared to the same frequencies at 6 months (the end of the intervention period). Better outcomes will be the same or lower frequencies of AYA concerns and symptoms at 9 months, as compared to the 6-month assessment point.
Quality of Life (QOL) | Up to 9 months
  Determine the Sustainability of the effects of YES on participants' quality of life, as measured by the generic (range: 31-143) and cancer-specific (range: 16-99) summary scores of the Quality of Life in Adult Cancer Survivors scale, from month 6 to month 9. Sustainability will be determined by both subscale scores maintaining the same or lower scores at 9 months as compared to their respective scores at month 6.

OTHER OUTCOMES:
Potential effects of the intervention on inflammatory and other biomarkers and genetic profiles | Baseline and 6 months
  We will measure pro- and anti-inflammatory cytokines (IL1β, IL6, IL8, IL10, TNF- α, and CRP) from participants' blood samples. We will also evaluate pro-inflammatory cytokine genes using microarray-based genome-wide transcriptional profiling to identify genes that show differential expression in leukocytes, aiming to accurately identify activation of specific transcription control pathways, including the pro-inflammatory NF-kB and decreased GR signaling. These pathways are hypothesized to underlie increased inflammatory activity, which may be more sensitive to our intervention than circulating cytokines, with improved symptom control and improved quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Naughton, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dibble KE, Rosenberg SM, Snow C, Kirkner GJ, Tayob N, Contreras M, Roma ND, DeGraffinreid CR, Nolan TS, Hershman DL, Naughton M, Partridge AH. Young, Empowered & strong (YES): a study protocol paper for a randomized controlled trial of an mHealth symptom monitoring and self-management intervention for adolescent and young adult (AYA) breast cancer survivors. BMC Public Health. 2025 Jan 11;25(1):126. doi: 10.1186/s12889-025-21288-4. PMID 39799291
- See also: The Jamesline — http://cancer.osu.edu